CLINICAL TRIAL: NCT07292649
Title: Maternal Expectations on Labor Analgesia and Risk of Postpartum Depression: An Observational Study
Status: Not yet recruiting | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Alessandro De Cassai, Principal Investigator, University of Padova
Other Study IDs: 6311/AO/25; AOP 3794 (Other: University Hospital of Padua, Italy)
Record Dates: First submitted 2025-09-13; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Postpartum Depression (PPD); Labor Analgesia; Expectations
Keywords: postpartum depression; labor analgesia; epidural; expectations
MeSH Terms: conditions — Depression, Postpartum | interventions — Analgesia, Epidural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Expectations met (Intended = Received): Participants whose prenatal intention regarding labor analgesia matched what they received (includes Intention Yes/Received Yes and Intention No/Received No).
  Interventions: Procedure: Epidural analgesia; Procedure: Spinal analgesia for labour pain; Other: No neuraxial analgesia
- Expectations unmet (Intended ≠ Received): Participants whose prenatal intention did not match the analgesia actually received (includes Intention Yes/Received No and Intention No/Received Yes).
  Interventions: Procedure: Epidural analgesia; Procedure: Spinal analgesia for labour pain; Other: No neuraxial analgesia

INTERVENTIONS:
Procedure: Epidural analgesia — Analgesia via epidural catheter using local anesthetic ± opioid, administered on patient request during labor.
Procedure: Spinal analgesia for labour pain — Single-shot spinal analgesia
Other: No neuraxial analgesia — Patients did not received spinal or epidural labour analgesia

SUMMARY:
Postpartum Depression (PPD) is defined as the development of depression at any time during the first year after childbirth¹. Its prevalence ranges from 15% to 20%. It can manifest with symptoms such as depressed mood, loss of interest and energy, insomnia, anxiety, and may even lead to suicidal ideation. The consequences are numerous, both physical and psychological, with long-term repercussions on the mother-infant bond, family dysfunction, and the development of emotional and cognitive disorders in children. The etiology of PPD is multifactorial, but numerous recent studies have focused on the role of labor pain and its management with labor analgesia techniques. The aim of the present study is therefore to assess whether there is a difference in the incidence of PPD between parturients whose expectations regarding labor analgesia were met ('expectations met' group) versus those whose expectations were unmet.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Planned vaginal delivery (spontaneous or induced)
* Pregnancy
* Age > 18 years

Exclusion Criteria:

* Allergy to local anesthetics
* Language barrier
* Contraindications to labor analgesia
* Delivery by Cesarean section
* Known history of psychiatric disorders (including major depression)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients undergoing a spontaneous or induced vaginal delivery, regardless of whether they request epidural analgesia.
Sampling Method: Non-Probability Sample
Enrollment: 3640 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
incidence of postpartum depression | 6 months since labour
  To assess whether there is a statistically significant difference in the incidence of postpartum depression (PPD), defined as an Edinburgh Postnatal Depression Scale (EPDS) score ≥ 10 at 6 months postpartum, between parturients whose expectations regarding labor analgesia were met ('expectations met' group) versus those whose expectations were unmet.

SECONDARY OUTCOMES:
Early depressive symptoms | from 24 to 48 hours since labour
  To assess whether there is a statistically significant difference in the incidence of postpartum depression (PPD), defined as an Edinburgh Postnatal Depression Scale (EPDS) score ≥ 10 at 6 months postpartum, between parturients whose expectations regarding labor analgesia were met ('expectations met' group) versus those whose expectations were unmet.
Effect of Analgesia Within Expectations-Unmet Group | six months since labour
  To compare the incidence of postpartum depression (EPDS ≥ 10 at 6 months) within the "Expectations unmet" group, stratified by actual receipt of neuraxial labor analgesia (epidural or spinal) versus no neuraxial analgesia
Pain Intensity and Maternal Expectations | At delivery/birth
  To assess the association between intrapartum pain intensity (measured by Visual Analog Scale, VAS) and group allocation ("Expectations met" vs "Expectations unmet").

IPD SHARING:
Plan to Share IPD: No